CLINICAL TRIAL: NCT03757975
Title: Impact of Hysterectomy and Supracervical Hysterectomy on Quality of Life, Urinary Incontinence and Urethral Length
Brief Title: Impact of Hysterectomy on Quality of Life and Urethral Length
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Paweł Miotła, Clinical Professor, Medical University of Lublin
Other Study IDs: 012018
Record Dates: First submitted 2018-11-19; First posted 2018-11-29 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Fibroid Uterus; Urethral Diseases; Sex Disorder
Keywords: quality of life; urethral length; sexual function
MeSH Terms: conditions — Leiomyoma; Urethral Diseases; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- TAH: patients before and after total abdominal hysterectomy (TAH)
  Interventions: Procedure: urethral length measure
- TLH: patients before and after total laparoscopic hysterectomy (TLH)
  Interventions: Procedure: urethral length measure
- TVH: patients before and after total vaginal hysterectomy (TVH)
  Interventions: Procedure: urethral length measure
- SAH: patients before and after abdominal supracervical hysterectomy (SAH)
  Interventions: Procedure: urethral length measure
- SLH: patients before and after supracervical laparoscopic hysterectomy (SLH)
  Interventions: Procedure: urethral length measure

INTERVENTIONS:
Procedure: urethral length measure — measure of urethral length, distribution of questionnaires before and after operation
  Other Names: UDI 6 and IIQ 7 questionnaires; FSFI questionnaire; ICIQ questionnaire

SUMMARY:
To establish the impact of hysterectomy on sexual function, urethral length and quality of life

DETAILED DESCRIPTION:
The investigators evaluate impact of total hysterectomy (abdominal, by laparoscopy and vaginal) and supracervical hysterectomy (abdominal and by laparoscopy) on quality of life, sexual function, urethral length and urinary incontinence. The patients fulfill questionnaires (UDI 6, IIQ7, FSFI and ICIQ) before operation and 6 months after. Additionally the investigators measure urethral length before procedure and 6 months after.

ELIGIBILITY:
Inclusion Criteria:

* patients qualified to hysterectomy due to benign condition

Exclusion Criteria:

* serious health condition
* previous vaginal operations

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women who have been qualified to hysterectomy due to fibroids or other benign cndition and who had not undergone any vaginal operation in the past
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline urethral length at 6 months after hysterectomy | 6 months
  Comparison of urethral length before and after hysterectomy. Urethra will be measured during ultrasound examination in millimeters

SECONDARY OUTCOMES:
Change from Baseline in sexual functions at 6 months after hysterectomy | 6 months
  The patients fulfill FSFI questionnaire before and after hysterectomy. Range 2-36 with higher scores indicating better sexual function.
Change from Baseline in appearance of urinary incontinence at 6 months after hysterectomy | 6 months
  The patients fulfill UDI 6 (range 0-400) questionnaire to assess appearance of urinary incontinence before and after hysterectomy
Change from Baseline in impact of urinary incontinence at 6 months after hysterectomy | 6 months
  The patients fulfill IIQ 7 (range 0-400) questionnaire to assess impact of hysterectomy on urinary incontinence.
Change from Baseline in urinary tract symptoms at 6 months after hysterectomy | 6 months
  The patients fulfill ICIQ questionnaire to assess impact of hysterectomy on urinary tract symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Rechberger, Professor, Study Director — Medical University of Lublin
Locations (1):
- 2nd Gynecology Department, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No